CLINICAL TRIAL: NCT06692868
Title: Fertility Protection for Children, Adolescents and Young Adults
Acronym: FeProCAYA
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Martin Wabitsch, Pediatric endocrinologist, University of Ulm
Other Study IDs: FeProCAYA
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Stem Cell Transplant; Stem Cell Transplantation; Oncological Outcomes; Oncological Patients; Oncological Children; Fertility; Fertility Protection; Endocrinological Late-effects; Paediatric Oncology; CAYA; Survivors
Keywords: FeProCAYA; Fertility protection; Endocrinological follow-up after oncological disease; children; fertility; adolescents; young adults; TYA; teenagers and young adults; paediatric oncology; follow-up care; endocrinological late-effects; survivors; stem cell transplant; stem cell transplantation; CAYA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Preservation of DNA and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- FeProCAYA-Onc: Children, adolescents, young adults (age <21 years) with a diagnosis of cancer before the initiation of oncological therapy or prior to SCT (stem cell transplantation) for a malignant or non-malignant disease with prospective follow-up.
- FeProCAYA-Onc (MidTerm): Children, adolescents, and young adults with a diagnosis of cancer before the age of 21 years and >5 years of follow-up after initial cancer diagnosis
- FeProCAYA-Onc (long-term): Adults with a diagnosis of cancer before the age of 21 years and >20 years of follow-up after initial cancer diagnosis
- FeProCAYA-SCT: Children and adolescents (age <21 years) with a malignant or non-malignant condition requiring stem cell transplantation (SCT) prior to SCT with prospective follow-up.

SUMMARY:
This study focuses on improving fertility preservation and long-term care for children, adolescents, and young adults (CAYA) undergoing cancer treatments or stem cell transplantation. These treatments can harm fertility, and ensuring that patients receive the right support and follow-up care is critical.

The main study goals are:

1. Understanding Fertility Risks: Researchers aim to identify factors that predict fertility problems after cancer treatments, such as the type of therapy, hormone levels, body composition, or genetic predispositions.
2. Addressing Patient and Family Needs: The program will explore the concerns, needs, and challenges faced by young patients and their parents regarding fertility. It will also examine how these issues affect their quality of life.
3. Improving Clinical Care: Current practices in fertility preservation and counseling will be studied to identify gaps and improve care structures.

To achieve these goals, the program will:

* Create a database to collect and analyze medical data from patients before, during, and after cancer treatments.
* Study the prevalence and long-term effects of fertility problems in young patients.
* Document medical interventions like fertility preservation methods (e.g., freezing eggs or sperm) and treatments for late effects.
* Assess patients' and families' fertility-related quality of life and their informational needs.

Ultimately, the project aims to establish an interdisciplinary center to support fertility preservation and improve the quality of care for young patients facing cancer and its treatments.

DETAILED DESCRIPTION:
The protection and preservation of fertility is particularly important for patients with tumor diseases prior to cell-damaging therapies, especially in pediatric oncology and during stem cell transplantation.

Fertility preservation in CAYA (Children, Adolescents, and Young Adults) remains a topic that receives limited attention in everyday clinical practice. While it has been addressed in pediatric oncology for years, it is often inconsistently implemented in daily ward routines and rarely adheres to clinical guidelines.

A rational strategy for fertility-preserving and endocrinological follow-up care should consider not only the therapeutic modalities employed in light of the patient's underlying disease but also the age and gender of the patient at the time of therapy.

The structured documentation of critical risk factors for the manifestation of fertility-restricting endocrinological late effects, as well as precise longitudinal documentation, are therefore of immediate importance in clinical patient care. They ensure the quality of diagnostic and therapeutic processes and outcomes and enable both retrospective and prospective scientific investigations.

The following key questions are central to this effort:

1. Can predictive factors or combined predictor variables for fertility disorders during follow-up be developed based on detailed clinical and laboratory phenotyping of patients before and after exposure to gonadotoxic therapies (e.g., therapeutic exposures, endocrinological markers, anthropometric markers such as body composition, genetic predispositions including risk SNPs and epigenetics)?
2. What unmet needs, concerns, and challenges regarding potential fertility impairments exist in different CAYA age groups and their parents, and how do these unmet needs affect the fertility-related quality of life of those affected?
3. How can current practices in fertility preservation and counseling for fertility preservation be systematically captured, with the goal of improving clinical care structures (healthcare research)?

These research questions will be addressed within the framework of a multimodal research program, specifically through:

1. Development and implementation of a database for the structured collection of therapy-related endocrinological, anthropometric, and laboratory parameters of patients before and after oncological therapy (or stem cell transplantation), as well as during follow-up care at the Department of Pediatrics and Adolescent Medicine, University Medical Center Ulm, Germany.
2. Identification of predictors for fertility disorders:

   1. Therapeutic exposures during primary and secondary therapy
   2. Endocrinological markers
   3. Anthropometric markers (body composition)
   4. Genetic predispositions
3. Prospective evaluation of the prevalence and cumulative incidence of fertility disorders in boys and girls during childhood and adolescence, including endocrinological and metabolic late effects.
4. Documentation of medical interventions, such as fertility-preserving measures before therapy, endocrinological treatments for late effects, and reproductive medical measures to support future parenthood (e.g., ICSI, IVF, IUI, oocyte transfer, etc.).
5. Assessment of previous fertility-preservation measures and counseling efforts for fertility preservation. The long-term goal is to improve the quality of patient care in endocrinological follow-up, focusing on fertility-related parameters after oncological diseases through the structured collection of relevant data.
6. Evaluation of fertility-related quality of life and informational needs at different time points during the course of the disease.

FeProCAYA is a part of the collaborative research project FePro-Ulm (https://www.uniklinik-ulm.de/frauenheilkunde-und-geburtshilfe/schwerpunkte/unifee/standard-titel.html), which is funded by the German Federal Ministry of Education and Research (BMBF). FePro-Ulm is an interdisciplinary junior scientists research center for fertility protection and one of five German CERES Excellence Centers for reproductive health (https://www.gesundheitsforschung-bmbf.de/de/interdisziplinaere-nachwuchszentren-fuer-reproduktive-gesundheit-16739.php).

ELIGIBILITY:
Children, adolescents, young adults with a diagnosis of cancer before the age of 21 years

or

Children, adolescents, young adults undergoing SCT for a malignant or non-malignant condition before the age of 21 years

treated at the Department of Pediatrics and Adolescent Medicine, University Medical Center Ulm, Germany.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mono-centric, prospective cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2044-11 (Estimated); Study Completion 2044-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence and cumulative incidence of endocrine sequelae of cancer treatments and SCT during childhood | 0 - >20 years after diagnosis or start of therapy
  Prospective evaluation of the prevalence and cumulative incidence of fertility disorders, including endocrinological and metabolic late effects, in childhood cancer survivors and children and adolescents who underwent SCT for malignant and non-malignant conditions during long-term follow-up care.
Predictors for fertility disorders in childhood cancer and SCT survivors | 0 - >20 years after diagnosis or start of therapy
  Identification of predictors for fertility disorders in childhood cancer survivors and patients, who underwent SCT during childhood, including:
  * Therapeutic exposures during primary and secondary therapy,
  * Endocrinological markers,
  * Anthropometric markers (e.g., body composition),
  * Genetic predisposition.

SECONDARY OUTCOMES:
Assessment of fertility-related quality of life | 0 - >20 years after diagnosis or start of therapy
  Structured and standardized assessment of fertility-related quality of life and informational needs at various time points throughout long-term follow-up care.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Denzer, Prof. Dr., Principal Investigator — Ulm University Medical Centre - Division of Paediatric Endocrinology and Diabetes; Martin Wabitsch, Prof. Dr., Study Chair — Ulm University Medical Centre - Division of Paediatric Endocrinology and Diabetes
Locations (1):
- Universitätsklinikum Ulm, Klinik für Kinder- und Jugendmedizin, Sektion Pädiatrische Endokrinologie und Diabetologie, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Project overview and information resources on research program and work packages (in German) — https://www.uniklinik-ulm.de/frauenheilkunde-und-geburtshilfe/schwerpunkte/unifee/standard-titel.html